CLINICAL TRIAL: NCT00346606
Title: A Randomized, Double-Blind, Active-Controlled, Parallel-Group Study to Compare the Efficacy and Safety of Desloratadine 5mg (Denosin®) With Levocetirizine 5mg (Xyzal®) in the Treatment of Chronic Idiopathic Urticaria Patients
Brief Title: The Efficacy and Safety of Desloratadine With Levocetirizine in Treatment of Chronic Idiopathic Urticaria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lotus Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 187CL1
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2006-06-30 (Estimated); Status verified 2006-05

CONDITIONS: Chronic Idiopathic Urticaria; Urticaria
Keywords: Chronic Idiopathic Urticaria; Desloratadine; Denosin; Levocetirizine
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — levocetirizine

INTERVENTIONS:
Drug: Denosin® and Xyzal®

SUMMARY:
Objective: To compare the efficacy of desloratadine 5mg (Denosin®) and levocetirizine 5mg (Xyzal®) once daily in the treatment of patients with CIU over 6 weeks.

Trial design: Randomized, Double-Blind, Active-Controlled, Parallel-Group Study.

Primary end point: To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the subjects' diaries during the first two weeks of the treatment.

Secondary Objectives: To assess the efficacy and safety of desloratadine 5mg (Denosin®) and levocetirizine 5mg (Xyzal®) once daily in the treatment of subjects with CIU over 6 weeks.

DETAILED DESCRIPTION:
Objective: To compare the efficacy of desloratadine 5mg (Denosin®) and levocetirizine 5mg (Xyzal®) once daily in the treatment of patients with CIU over 6 weeks.

Trial design: Randomized, Double-Blind, Active-Controlled, Parallel-Group Study.

Primary endpoint: To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the subjects' diaries during the first two weeks of the treatment.

Secondary Objectives: To assess the efficacy and safety of desloratadine 5mg (Denosin®) and levocetirizine 5mg (Xyzal®) once daily in the treatment of subjects with CIU over 6 weeks.

Primary endpoint:

To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the patient diaries during the first two weeks of treatment

Secondary Endpoints- To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the subjects' diaries over the 6 weeks.

To evaluate the reflective average AM/PM scores for number of hives, size of largest hive, and total symptom score (sum of pruritus, number of hives, and size of largest hive scores).

Average individual AM/PM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.

AM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.

PM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.

PM reflective scores for pruritus, number of hives, and size of largest hive are also evaluated.

The interference with sleep (AM reflective), and interference with daily activities (PM reflective) are other secondary efficacy outcomes.

Therapeutic response will be evaluated at visit 3~5.

Safety will be evaluated including vital signs are recorded at all visits, whereas sleep latency using Epworth Sleepiness Scale (ESS) questionnaire and Visual analogue Scale (VAS) are scored at visit 2~5. Stanford Sleepiness Scale (SSS) are scored according to the instructions of diary cards at all visits. All adverse events are recorded and graded for severity at visit 2~5.

ELIGIBILITY:
Inclusion Criteria:

* The subject or deputy has read or been informed and signed the Informed Consent Agreement and the subject will be willing and able to participate in the study.
* The subject ≥ 12 years old.
* The subject with documented signs and symptoms of CIU for 6 weeks or more.
* The subject has to have a CIU flare for 3 weeks or more before screening, with urticarial lesions visible 3 days or more per week.
* The overall severities of CIU have to be at least mild to moderate at screening and baseline, subjects have to have at least mild to moderate pruritus, hives have to be apparent at screening, and subjects have intention to treatment.

Exclusion Criteria:

* The subject has received any histamine, corticosteroids, ketotifene, systemic antibiotics, nedocromil, sodium cromoglycate or thyroxin drug within 7 days preceding randomization.
* The subject has received any other investigational drug within one month preceding randomization.
* The subject has previous non-response to antihistamines.
* The subject has previous allergy or allergies of desloratadine or levocetirizine.
* The subject need for long-term corticosteroids treatment (including inhaled, oral and topical dosage).
* The subject has autoimmune diseases.
* The subject's urticaria is physical urticaria, cholinergic urticaria or angioedema.
* The subject is in the situation of pregnancy or breastfeeding.
* The subject has liver dysfunction (AST ≧ 3 times normal range; ALT ≧ 3 times normal range ) or renal dysfunction (Creatinine ≧ 3.0mg/dl ).
* The subject is unable to keep an accurate diary of disease symptoms.
* The subject has significant concomitant illness, which, in the opinion of the investigator, will interfere with the evaluation of the study medications.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01

PRIMARY OUTCOMES:
To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the patient diaries during the first two weeks of treatment

SECONDARY OUTCOMES:
To evaluate the change in average AM/PM reflective pruritus score from baseline recorded in the subjects' diaries over the 6 weeks.
To evaluate the reflective average AM/PM scores for number of hives, size of largest hive, and total symptom score (sum of pruritus, number of hives, and size of largest hive scores).
Average individual AM/PM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.
AM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.
PM instantaneous scores for pruritus, number of hives, and size of largest hive are also evaluated.
PM reflective scores for pruritus, number of hives, and size of largest hive are also evaluated.
The interference with sleep (AM reflective), and interference with daily activities (PM reflective) are other secondary efficacy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Yu Chu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Dermatology National Taiwan University Hospital, Taipei, Taiwan